CLINICAL TRIAL: NCT04674098
Title: The Effect of Real Time Analytics on Adverse Events Among Hospitalized Patients
Status: Withdrawn | Type: Observational
Why Stopped: COVID protocols limited access to data. PI then moved to a different institution
Sponsor: Bob Topp (Other)
Responsible Party: Sponsor-Investigator, Bob Topp, Professor, University of Toledo
Organization: University of Toledo (Other)
Other Study IDs: 300854-UT
Record Dates: First submitted 2020-12-04; First posted 2020-12-19 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Hospital Acquired Condition
MeSH Terms: conditions — Iatrogenic Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

GROUPS / COHORTS (2):
- Usual Care: Every patient who is admitted or transferred to the target unit during both the baseline and intervention phases of the study will be approached by a member of the research staff to be a subject in the study. The patient will be informed of the overall study objectives and be requested to provide informed consent to participate. The patient's involvement in the study will include having the research staff access and extract relevant outcome variables collected from their electronic health record (EHR) (AEs, admissions to the ICU, hospital length of stay and activation of the rapid response team) as a result of their hospital stay.
- Intervention: If the patient provides consent during the intervention phase, the BAS technology will passively monitor their vital signs generated by the Philips vital sign monitor by relaying their deidentified vital signs data to the CLU, proprietary Cloud server, and subsequently Lumori® on a study-issued cell phone of the RN who is primarily responsible for the patient's care. Patient's admitted or transferred to the targeted unit will NOT be excluded from being approached to participate in the study.
  Interventions: Device: The Beat Analytics System (BAS)

INTERVENTIONS:
Device: The Beat Analytics System (BAS) — There are three subsystems to the BAS; data aggregation, data analysis and data presentation.
  Groups: Intervention

SUMMARY:
This study will examine the effect of providing nurses with continuous, remote, real-time monitoring of their patient's vital signs and MEWS scores using the BAS on the occurrence of adverse events, admissions to the ICU, hospital length of stay and activation of the rapid response team among patients on non-intensive care hospital units. A longitudinal study will measure the outcome variables among an estimated 60 patients per month during 6 month intervals when the BAS is not and is available to the nursing staff.

DETAILED DESCRIPTION:
Adverse events (AEs) among hospitalized patients are defined as "Unintended injuries or complications that result in disability at discharge, death or prolonged hospital stay and are caused by events other than the patient's underlying disease." Annually, approximately 1.1% of all hospital admissions, or 400,000 patients, die due to AEs while costing the US economy roughly 17.1 billion dollars. The Canadian Adverse Events Study reported AEs among 7.5% of hospital admissions, with 37% of these events deemed preventable. Common AEs, including infections and sepsis, cardiac and respiratory failure and deaths have been reported to be proceeded by a change in the patient's vital signs recognizable up to 48 hours prior to the AE being diagnosed. In many cases, subtle changes in a patient's vital signs have been recognized retrospectively as precursors of AEs that can lead to unplanned admissions to ICUs or death.

A number of early warning systems have been developed to assist nursing staff in identifying changes in vital signs as precursors to AEs. The commonly used Modified Early Warning Score (MEWS) attempts to identify acute clinical deterioration based on the patient's vital signs and level of consciousness. The higher the MEWS score, the greater risk of an AE. However, the efficacy of the MEWS score is contingent upon the frequency of both the score being recorded and being assessed by the nursing staff. Although continuous monitoring of vital signs takes place within and outside of ICUs these data are rarely provided to the nurse when they are outside of the patient's room in real time. Further, the vital signs and MEWS scores are commonly recorded in the patient record at scheduled intervals during a 24-hour period (e.g. every 4, 6, 8 or 12 hours). If a patient's physiological condition deteriorates between these scheduled intervals and the nurse is not continually with the patient, the opportunity is lost for early recognition of this deterioration that may lead to an AE. The importance of monitoring vital signs in clinical practice is indisputable, but how to best monitor and interpret them and how frequently they should be measured in order to minimize AEs remains unclear.

In order to address this gap in the literature, the project team has developed an innovative technology. The Beat Analytics System (BAS) provides nurses with both real-time monitoring of the patient's vital signs and continuous calculation of their patient's MEWS scores through an app on their cell phone. This information can be presented both numerically (with boundary conditions for alerts) and graphically, in order to observe change in the MEWS score over time. The purpose of this study is to examine the effect of providing nurses with remote, continuous, real-time monitoring of their patients vital signs and MEWS scores using the BAS on the occurrence of AEs, admissions to the ICU, hospital length of stay, and activation of the rapid response team among patients on non-intensive care hospital units. This purpose will be addressed through a longitudinal sequential study design in which the outcome variables (AEs, admissions to the ICU hospital length of stay and activation of the rapid response team) will be monitored on two 20-bed non-intensive care units monthly for 6 months without the BAS. The 6-month baseline data collection period will be followed by a month of training the nursing staff on the targeted unit to using the BAS. Following this orientation month, the outcome variables will again be measured during a 6-month intervention phase in which the BAS will be available to the nurses caring for patients on the targeted unit where the patient's vital signs will be continually recorded.

ELIGIBILITY:
Inclusion Criteria:

* Admitted to one of two non-intensive care units within the University of Toledo Medical Center (UTMC) hospital.

Exclusion Criteria:

* unable to provide informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects for this study will include patients who are admitted to one of the two non-intensive care targeted units within the UTMC hospital.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Adverse events | during hospital admission averaging 7 days
  Development of an infection or sepsis, cardiac or respiratory failure, and death
Length of stay in the hospital | during hospital admission averaging 7 days
  Duration of days during which a subject was admitted to the hospital
Transfer to the ICU | during hospital admission averaging 7 days
  Transfer of the patient to the intensive care unit
RRT activation | during hospital admission averaging 7 days
  Activation of the hospital's rapid response team to support the care of the patient

CONTACTS AND LOCATIONS:
Overall Officials: Robert Topp, PhD, Principal Investigator — College of Nursing
Locations (1):
- The University of Toledo Medical Center, Toledo, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
No Plan Has been developed

REFERENCES:
- [Result] Unbeck M, Schildmeijer K, Henriksson P, Jurgensen U, Muren O, Nilsson L, Pukk Harenstam K. Is detection of adverse events affected by record review methodology? an evaluation of the "Harvard Medical Practice Study" method and the "Global Trigger Tool". Patient Saf Surg. 2013 Apr 15;7(1):10. doi: 10.1186/1754-9493-7-10. PMID 23587448
- [Result] Van Den Bos J, Rustagi K, Gray T, Halford M, Ziemkiewicz E, Shreve J. The $17.1 billion problem: the annual cost of measurable medical errors. Health Aff (Millwood). 2011 Apr;30(4):596-603. doi: 10.1377/hlthaff.2011.0084. PMID 21471478
- [Result] Lapointe-Shaw L, Bell CM. Measuring the cost of adverse events in hospital. CMAJ. 2019 Aug 12;191(32):E877-E878. doi: 10.1503/cmaj.190912. No abstract available. PMID 31613792
- [Result] Islam MM, Nasrin T, Walther BA, Wu CC, Yang HC, Li YC. Prediction of sepsis patients using machine learning approach: A meta-analysis. Comput Methods Programs Biomed. 2019 Mar;170:1-9. doi: 10.1016/j.cmpb.2018.12.027. Epub 2018 Dec 26. PMID 30712598
- [Result] Kim J, Chae M, Chang HJ, Kim YA, Park E. Predicting Cardiac Arrest and Respiratory Failure Using Feasible Artificial Intelligence with Simple Trajectories of Patient Data. J Clin Med. 2019 Aug 29;8(9):1336. doi: 10.3390/jcm8091336. PMID 31470543
- [Result] Jayasundera R, Neilly M, Smith TO, Myint PK. Are Early Warning Scores Useful Predictors for Mortality and Morbidity in Hospitalised Acutely Unwell Older Patients? A Systematic Review. J Clin Med. 2018 Sep 28;7(10):309. doi: 10.3390/jcm7100309. PMID 30274205
- [Result] Kause J, Smith G, Prytherch D, Parr M, Flabouris A, Hillman K; Intensive Care Society (UK); Australian and New Zealand Intensive Care Society Clinical Trials Group. A comparison of antecedents to cardiac arrests, deaths and emergency intensive care admissions in Australia and New Zealand, and the United Kingdom--the ACADEMIA study. Resuscitation. 2004 Sep;62(3):275-82. doi: 10.1016/j.resuscitation.2004.05.016. PMID 15325446
- [Result] Downey CL, Tahir W, Randell R, Brown JM, Jayne DG. Strengths and limitations of early warning scores: A systematic review and narrative synthesis. Int J Nurs Stud. 2017 Nov;76:106-119. doi: 10.1016/j.ijnurstu.2017.09.003. Epub 2017 Sep 13. PMID 28950188
- [Result] Ludikhuize J, Smorenburg SM, de Rooij SE, de Jonge E. Identification of deteriorating patients on general wards; measurement of vital parameters and potential effectiveness of the Modified Early Warning Score. J Crit Care. 2012 Aug;27(4):424.e7-13. doi: 10.1016/j.jcrc.2012.01.003. Epub 2012 Feb 14. PMID 22341727
- [Result] Kim WY, Shin YJ, Lee JM, Huh JW, Koh Y, Lim CM, Hong SB. Modified Early Warning Score Changes Prior to Cardiac Arrest in General Wards. PLoS One. 2015 Jun 22;10(6):e0130523. doi: 10.1371/journal.pone.0130523. eCollection 2015. PMID 26098429
- [Result] van Galen LS, Dijkstra CC, Ludikhuize J, Kramer MH, Nanayakkara PW. A Protocolised Once a Day Modified Early Warning Score (MEWS) Measurement Is an Appropriate Screening Tool for Major Adverse Events in a General Hospital Population. PLoS One. 2016 Aug 5;11(8):e0160811. doi: 10.1371/journal.pone.0160811. eCollection 2016. PMID 27494719
- [Result] Wang AY, Fang CC, Chen SC, Tsai SH, Kao WF. Periarrest Modified Early Warning Score (MEWS) predicts the outcome of in-hospital cardiac arrest. J Formos Med Assoc. 2016 Feb;115(2):76-82. doi: 10.1016/j.jfma.2015.10.016. Epub 2015 Dec 24. PMID 26723861
- [Result] Brekke IJ, Puntervoll LH, Pedersen PB, Kellett J, Brabrand M. The value of vital sign trends in predicting and monitoring clinical deterioration: A systematic review. PLoS One. 2019 Jan 15;14(1):e0210875. doi: 10.1371/journal.pone.0210875. eCollection 2019. PMID 30645637
- [Result] Smith GB, Recio-Saucedo A, Griffiths P. The measurement frequency and completeness of vital signs in general hospital wards: An evidence free zone? Int J Nurs Stud. 2017 Sep;74:A1-A4. doi: 10.1016/j.ijnurstu.2017.07.001. Epub 2017 Jul 4. No abstract available. PMID 28701265
- [Result] Yoder JC, Yuen TC, Churpek MM, Arora VM, Edelson DP. A prospective study of nighttime vital sign monitoring frequency and risk of clinical deterioration. JAMA Intern Med. 2013 Sep 9;173(16):1554-5. doi: 10.1001/jamainternmed.2013.7791. No abstract available. PMID 23817602